CLINICAL TRIAL: NCT01300546
Title: TreximetTM in the Prevention and Modification of Disease Progression in Migraine
Brief Title: Treximet Trademark (TM) in the Prevention and Modification of Disease Progression in Migraine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cady, Roger, M.D. (Individual)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 114933
Record Dates: First submitted 2011-01-12; First posted 2011-02-21 (Estimated); Results first posted 2013-05-21 (Estimated); Last update posted 2013-05-21 (Estimated); Status verified 2013-05

CONDITIONS: Migraine
Keywords: Frequent migraine; Migraine transformation; Migraine; Treximet; Naproxen; Sumatriptan
MeSH Terms: conditions — Migraine Disorders | interventions — Sumatriptan; Naproxen; sumatriptan-naproxen

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sumatriptan/Naproxen Sodium (Active Comparator): In Treatment Period, subjects randomized to Sumatriptan/Naproxen Sodium will be provided with 14 tablets of Sumatriptan/Naproxen Sodium to treat migraine within 1 hour of onset on 14 or fewer days per month. Subjects will be provided with 14 tablets of Sumatriptan/Naproxen Sodium per month for rescue of persistent or recurring headache.
  Interventions: Drug: Sumatriptan/Naproxen Sodium
- Naproxen Sodium (Active Comparator): In Treatment Period, subjects randomized to Naproxen Sodium 500mg will be provided with 14 tablets of Naproxen Sodium to treat migraine within 1 hour of onset on 14 or fewer days per month. Subjects will be provided with 14 tablets of Naproxen Sodium per month for rescue of persistent or recurring headache.
  Interventions: Drug: Naproxen Sodium

INTERVENTIONS:
Drug: Sumatriptan/Naproxen Sodium — Each tablet of Treximet for oral administration contains Sumatriptan 85mg / Naproxen Sodium 500mg. Study medication is to be administered within 1 hour of migraine onset on 14 or fewer days per month in the Treatment Period.
  Other Names: Treximet
  Arms: Sumatriptan/Naproxen Sodium
Drug: Naproxen Sodium — Each tablet of Naproxen Sodium for oral administration is provided in 500mg tablet. Study medication is to be administered within 1 hour of migraine onset on 14 or fewer days per month in the Treatment Period.
  Other Names: Naproxen
  Arms: Naproxen Sodium

SUMMARY:
This study is being conducted to evaluate the hypothesis that use of pharmacological and non-pharmacological interventions may allow subjects at high risk for chronic migraine to avoid or reverse the transformation of episodic migraine to chronic migraine.

DETAILED DESCRIPTION:
Two investigative centers will enroll 40 subjects in the United States. Subject participation in the 5 visit study will last 4 months.

At Visit 1, following informed consent, a medical, migraine, and medication history will be collected and a physical and neurological exam with vital signs will be performed. An electrocardiogram (ECG) will be completed. A Lifestyle Choices for Better Migraine Management Questionnaire (Lifestyle Questionnaire) will be completed. Eligible subjects then complete a 1-month Baseline Period and treat migraine with their current preferred treatment of choice, documenting headache severity and associated symptoms in a 30-day Baseline Diary.

At Visit 2, the Baseline Diary will be reviewed and a pregnancy test will be collected from all subjects of childbearing potential. Vital signs will be collected and Adverse Events documented. Subjects continuing to meet eligibility criteria will be randomized 1:1 to Treximet or naproxen and provided with study medication to treat on 14 or fewer days per month. Subjects will be encouraged to treat their migraine attacks within 1 hour of onset of headache pain and while the pain is still mild. Subjects will view an educational digital video disc (DVD) concerning lifestyle modification, receive a copy for home viewing, complete the Lifestyle Questionnaire, and receive 3 copies of the Lifestyle Questionnaire for weekly completion between Visits 2 and 3. The Migraine Disability Assessment questionnaire (MIDAS) will be completed and a 30-day Treatment Period Diary will be dispensed.

At Visits 3 and 4, Adverse Events will be collected, completed Diaries will be reviewed, and Drug Accountability performed. Pregnancy tests will be collected from all subjects of childbearing potential. Vital signs will be collected. Completed Lifestyle Questionnaires will be collected, a Lifestyle Questionnaire will be completed in the office, and 3 copies will be dispensed for weekly completion between visits. Study medication for the following month will be dispensed with a 30-day Diary.

At Visit 5, Adverse Events will be collected, completed Diaries will be reviewed, and Drug Accountability performed. Pregnancy tests will be collected from all subjects of childbearing potential. Vital signs will be collected. Completed Lifestyle Questionnaires will be collected and a Lifestyle Questionnaire will be completed in the office. Subjects will complete the MIDAS before exiting the study.

ELIGIBILITY:
Inclusion Criteria:

Subject

* Is male or female, in otherwise good health, 18 to 65 years of age.
* Has history of frequent episodic migraine (6-14 migraine days per month) (with or without aura) according to the 2nd Edition of The International Headache Classification (ICHD-2) for at least 3 months. (Stage 2-3 frequent transforming migraine)
* Had onset of migraine before age 50.
* Is able to differentiate migraine from any other headache they may experience (e.g., tension-type headache).
* Has stable history of headache at least 3 months prior to screening.
* Is not currently taking a migraine preventive or has been taking preventive for at least 30 days prior to screening and agrees to not start, stop, or change medication and/or dosage during the study period.
* Has at least 50% of migraine attacks beginning at mild severity.
* If female of childbearing potential, has a negative urine pregnancy test at Visits 1-5 and uses, or agrees to use, for the duration of the study, a medically acceptable form of contraception as determined by the investigator.

  1. Complete abstinence from intercourse from 2 weeks prior to administration of study drug throughout the study, and for a time interval after completion or premature discontinuation from the study to account for elimination of the study drug (a minimum of 7 days); or,
  2. Surgically sterile (hysterectomy or tubal ligation or otherwise incapable of pregnancy); or,
  3. Sterilization of male partner; or,
  4. Intrauterine device with published data showing lowest expected failure rate is less than 1% per year; or,
  5. Double barrier method (i.e., 2 physical barriers OR 1 physical barrier plus spermicide) for a least 1 month prior to Visit 1 and throughout study; or,
  6. Hormonal contraceptives for at least 3 months prior to Visit 1 and throughout study.
* Had 6 or more migraine treatment days in 1 month prior to Visit 2.

Exclusion Criteria:

Subject

* Is unable to understand the study requirements, the informed consent, or complete headache records as required per protocol.
* Is pregnant, actively trying to become pregnant, or breast-feeding.
* Has experienced the following migraine variants: basilar migraine, aura without headache, familial hemiplegic migraine, complicated migraine, ophthalmoplegic migraine and retinal migraine.
* Has a history of Medication Overuse Headache in the 3 months prior to study enrollment or during the baseline phase
* Has history of acute migraine treatment greater than14 days per month in 3 months prior to screening.
* Has abused, in the opinion of the Investigator, any of the following drugs, currently or within the past 1 year:

  1. opioids
  2. alcohol
  3. barbiturates
  4. benzodiazepine
  5. cocaine
* Has history of impaired hepatic or renal function that, in the investigator's opinion, contraindicates participation in this study.
* Has an unstable neurological condition or a significantly abnormal neurological examination with focal signs or signs of increased intracranial pressure.
* Suffers from cardiovascular disease (ischemic heart disease, including angina pectoris, myocardial infarction, documented silent ischemia, or with Prinzmetal's angina); has symptoms of ischemic heart disease, ischemic abdominal syndromes, peripheral vascular disease or Raynaud's Syndrome; has uncontrolled hypertension (≥140/90 millimeters of mercury (mmHg) in 2 out of 3 blood pressure (BP) measurements at screening); has electrocardiogram (ECG) results outside normal limits for clinically stable patients as judged by the investigator.
* Has a history of asthma and nasal polyps.
* Has a history of peptic ulcer disease requiring therapeutic intervention in the year prior to study enrollment
* Has evidence or history of any gastrointestinal (GI) surgery or GI ulceration or perforation of the stomach or intestine in the past 6 months, gastrointestinal bleeding in the past year or evidence or history of inflammatory bowel disease or history of any other bleeding disorder, or has taken or plans to take any anti-coagulant or any antiplatelet agent within the 2 weeks prior to screening through 48 hours post final study treatment.
* Has history of non-steroidal anti-inflammatory drug induced gastritis, esophagitis, or duodenitis.
* Suffers from a serious illness, or an unstable medical condition, one that could require hospitalization, or could increase the risk of adverse events.
* Has in the opinion of the investigator a significant cardiovascular risk profile that may include uncontrolled high blood pressure, post-menopausal women, male over 40 years old, hypercholesterolemia, obesity, diabetes mellitus, smoking, or a family history of cardiovascular disease in a 1st degree relative.
* Has in the opinion of the investigator a significant cerebrovascular risk profile that may include female over the age of 35 using oral birth control, smoking, or a family history of cerebrovascular disease in a first degree relative.
* Has a psychiatric condition, in the opinion of the investigator that may affect the interpretation of efficacy and safety data or contraindicates the subject's participation in the study.
* Has hypersensitivity, intolerance, or contraindication to the use of sumatriptan, any of its components, or any other 5-hydroxytryptamine 1 (5-HT1) agonist.
* Has a hypersensitivity, intolerance, or contraindication to the use of naproxen, any of its components, or any other non-steroidal anti-inflammatory drug including aspirin and cyclooxygenase-2 (COX-2) inhibiting agents.
* Is currently taking a migraine prophylactic medication containing an ergotamine or ergot derivative such as dihydroergotamine (DHE) or methysergide.
* Has taken, or plans to take, a monoamine oxidase inhibitor (MAOI) including herbal preparations containing St. John's wort (Hypericum perforatum), anytime within the 2 weeks prior to screening through 2 weeks post final study treatment.
* Has taken or plans to take an angiotensin-converting enzyme (ACE) inhibitor or angiotensin receptor blocker (ARB) anytime within the 2 weeks prior to screening through 48 hours post final study treatment.
* Has received any investigational agents within 30 days prior to Visit 1.
* Plans to participate in another clinical study at any time during this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2010-12; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roger K Cady, MD, Principal Investigator — Clinvest
Locations (2):
- United States (2):
  - Newport Beach Clinical Research Assoc., Inc., Newport Beach, California
  - Clinvest, Springfield, Missouri

REFERENCES:
- [Background] Cady RK, Goldstein J, Silberstein S, Juhasz M, Ramsey K, Rodgers A, Hustad CM, Ho T. Expanding access to triptans: assessment of clinical outcome. Headache. 2009 Nov-Dec;49(10):1402-13. doi: 10.1111/j.1526-4610.2009.01532.x. Epub 2009 Oct 8. PMID 19817885
- [Background] Cady RK, Martin VT, Geraud G, Rodgers A, Zhang Y, Ho AP, Hustad CM, Ho TP, Connor KM, Ramsey KE. Rizatriptan 10-mg ODT for early treatment of migraine and impact of migraine education on treatment response. Headache. 2009 May;49(5):687-96. doi: 10.1111/j.1526-4610.2009.01412.x. PMID 19472447
- [Background] Bigal ME, Sheftell FD, Rapoport AM, Lipton RB, Tepper SJ. Chronic daily headache in a tertiary care population: correlation between the International Headache Society diagnostic criteria and proposed revisions of criteria for chronic daily headache. Cephalalgia. 2002 Jul;22(6):432-8. doi: 10.1046/j.1468-2982.2002.00384.x. PMID 12133042
- [Background] Headache Classification Committee; Olesen J, Bousser MG, Diener HC, Dodick D, First M, Goadsby PJ, Gobel H, Lainez MJ, Lance JW, Lipton RB, Nappi G, Sakai F, Schoenen J, Silberstein SD, Steiner TJ. New appendix criteria open for a broader concept of chronic migraine. Cephalalgia. 2006 Jun;26(6):742-6. doi: 10.1111/j.1468-2982.2006.01172.x. PMID 16686915
- [Background] Lipton RB, Stewart WF, Cady R, Hall C, O'Quinn S, Kuhn T, Gutterman D. 2000 Wolfe Award. Sumatriptan for the range of headaches in migraine sufferers: results of the Spectrum Study. Headache. 2000 Nov-Dec;40(10):783-91. doi: 10.1046/j.1526-4610.2000.00143.x. PMID 11135021
- [Background] Newman LC, Lipton RB, Lay CL, Solomon S. A pilot study of oral sumatriptan as intermittent prophylaxis of menstruation-related migraine. Neurology. 1998 Jul;51(1):307-9. doi: 10.1212/wnl.51.1.307. PMID 9674831
- [Background] Foley KA, Cady R, Martin V, Adelman J, Diamond M, Bell CF, Dayno JM, Hu XH. Treating early versus treating mild: timing of migraine prescription medications among patients with diagnosed migraine. Headache. 2005 May;45(5):538-45. doi: 10.1111/j.1526-4610.2005.05107.x. PMID 15953272
- [Background] Rapoport AM, Bigal ME, Volcy M, Sheftell FD, Feleppa M, Tepper SJ. Naratriptan in the preventive treatment of refractory chronic migraine: a review of 27 cases. Headache. 2003 May;43(5):482-9. doi: 10.1046/j.1526-4610.2003.03094.x. PMID 12752754
- [Background] Sheftell FD, Rapoport AM, Tepper SJ, Bigal ME. Naratriptan in the preventive treatment of refractory transformed migraine: a prospective pilot study. Headache. 2005 Nov-Dec;45(10):1400-6. doi: 10.1111/j.1526-4610.2005.00273.x. PMID 16324173

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period was from date of Institutional Review Board (IRB) approval (11-30-10) until date last patient enrolled (1/3/12). Subjects were recruited from general population at two clinical research centers.
Pre-assignment Details: Subjects must complete a 30 day Baseline Period between Visit 1 and Visit 2 before Randomization. Subjects must have had 6-14 headache days during the 30 day Baseline Period in order to be Randomized into the Study Treatment Period. Fifty nine subjects were screened for study; however, only 39 subjects randomized for treatment due to screen fail.
Period: Overall Study
Arm/Group | Sumatriptan/Naproxen Sodium | Naproxen Sodium
Started | 19 | 20
Completed | 18 | 14
Not Completed | 1 | 6
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Lost to Follow-up | 0 | 2
Not completed — Lack of Efficacy | 0 | 3
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sumatriptan/Naproxen Sodium | Naproxen Sodium | Total
Number analyzed (Participants) | 19 | 20 | 39
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 19 | 20 | 39
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 35.7 (9.6) | 43.1 (9.3) | 39.5 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 19 | 36
  Male | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 19 | 20 | 39

OUTCOME MEASURES:

1. Primary Outcome: Percent Change of Headache Days Compared to Baseline
Description: Comparing the number of migraine headache days during Baseline Period Days 1-30 to number or migraine headache days reported in Treatment Period Days 91-120 in Sumatriptan/Naproxen Sodium arm vs. Naproxen Sodium arm. Percent change=[ (total headache days during Treatment Period Month 3 (Days 91-120)-total headache days during Baseline (Days 1-30)/total headache days during Baseline (Days 1-30)]*100%).
Time Frame: Day 121 (following 30 day Baseline Period and Treatment Period Days 91-120)
Measure: Mean (Standard Deviation); unit: percent change of headache days
Arm/Group | Sumatriptan/Naproxen Sodium | Naproxen Sodium
Number analyzed (Participants) | 18 | 14
percent change of headache days | -13.50 (34.80) | -36.50 (36.48)

2. Secondary Outcome: Migraine Attacks
Description: Comparing the number of migraine attacks reported from Baseline to the number of migraine attacks reported in Treatment Period Months 1(Days 31-60), 2(Days 61-90), and 3(Days 91-120) in Sumatriptan/Naproxen Sodium arm vs. Naproxen Sodium arm. Each treatment month percent change was individually compared to Baseline. The following formula was used for each treatment period calculation. e.g.,Percent change=[ (total migraine attacks days during Treatment Period Month 3 (Days 91-120)-total migraine attacks during Baseline (Days 1-30)/total migraine attacks during Baseline (Days 1-30)]*100%).
Time Frame: Baseline Period collected at Day 31, Treatment Period Months 1, 2, and 3 collected at Days 61, 91, and 121.
Measure: Mean (Standard Deviation); unit: percent change of migraine attacks
Arm/Group | Sumatriptan/Naproxen Sodium | Naproxen Sodium
Number analyzed (Participants) | 18 | 14
percent change of migraine attacks
  Baseline to Treatment Period Month 1 | -4.35 (32.63) | -12.23 (31.27)
  Baseline to Treatment Period Month 2 | -2.88 (37.59) | -9.03 (25.69)
  Baseline to Treatment Period Month 3 | -8.63 (38.10) | -39.12 (30.28)

3. Secondary Outcome: Migraine Severity
Description: Comparing migraine severity 2 hours after treatment from Baseline(Days 1-30) to migraine severity reported 2 hours after treatment in Treatment Period Months 1 (Days 31-60), 2(Days 61-90), and 3(Days 91-120) in Sumatriptan/Naproxen Sodium arm vs. Naproxen Sodium arm. Percent change was calculated by determining percent change in each subject, from Treatment Period Month 3 and Baseline, then comparing the average change between each arm. The following formula was used for each treatment period calculation. e.g.,Percent change=[ (mean migraine severity during Treatment Period Month 3 (Days 91-120)- mean migraine severity during Baseline (Days 1-30)/mean migraine severity during Baseline (Days 1-30)]*100%).
Time Frame: Baseline Period collected at Day 31, Treatment Period Months 1, 2, and 3 collected at Days 61, 91, and 121.
Measure: Mean (Standard Deviation); unit: percent change of migraine severity
Arm/Group | Sumatriptan/Naproxen Sodium | Naproxen Sodium
Number analyzed (Participants) | 18 | 14
percent change of migraine severity
  2 hours after treatment for Baseline to Month 1 | -17.84 (72.91) | 11.78 (79.60)
  2 hours after treatment for Baseline to Month 2 | -36.71 (49.78) | 0.33 (54.96)
  2 hours after treatment for Baseline to Month 3 | -55.60 (52.92) | 32.62 (107.62)

4. Secondary Outcome: Migraine Duration From Onset to Pain Free
Description: Comparing mean migraine duration from onset to painfree from Baseline(Days 1-30) to each month: Treatment Period Months 1 (Days 31-60), 2(Days 61-90), and 3(Days 91-120) in Sumatriptan/Naproxen Sodium arm vs. Naproxen Sodium arm. Percent change was calculated by determining percent change in each subject, from Treatment Period Month 3 and Baseline, then comparing the average change between each arm. The following formula was used for each treatment period calculation. e.g.,Percent change=[(mean duration from onset to painfree during Treatment Period Month 3 (Days 91-120)- mean duration from onset to painfree during Baseline (Days 1-30)/mean duration from onset to painfree during Baseline (Days 1-30)]*100%).
Time Frame: Baseline Period collected at Day 31, Treatment Period Months 1, 2, and 3 collected at Days 61, 91, and 121.
Measure: Mean (Standard Deviation); unit: percent change of migraine duration
Arm/Group | Sumatriptan/Naproxen Sodium | Naproxen Sodium
Number analyzed (Participants) | 18 | 14
percent change of migraine duration
  Baseline to Treatment Period Month 1 | 72.04 (214.89) | -14.92 (75.02)
  Baseline to Treatment Period Month 2 | 35.86 (178.63) | -26.35 (47.97)
  Baseline to Treatment Period Month 3 | 61.96 (304.74) | 70.84 (221.11)

5. Secondary Outcome: Migraine Duration From Time of Treatment to Pain Free
Description: % change from Baseline in mean migraine duration from time of treatment to pain free reported in Treatment Period Months 1, 2, and 3 in Sumatriptan/Naproxen Sodium arm vs. Naproxen Sodium arm.
  Percent change=[(mean duration from treatment to painfree during Treatment Period Month 3 (Days 91-120)- mean duration from treatment to painfree during Baseline (Days 1-30)/mean duration from treatment to painfree during Baseline (Days 1-30)]*100%).
Time Frame: Baseline Period collected at Day 31, Treatment Period Months 1, 2, and 3 collected at Days 61, 91, and 121.
Measure: Mean (Standard Deviation); unit: percent change of migraine duration
Arm/Group | Sumatriptan/Naproxen Sodium | Naproxen Sodium
Number analyzed (Participants) | 18 | 14
percent change of migraine duration
  Baseline to Treatment Period Month 1 | 150.10 (366.03) | -14.91 (76.85)
  Baseline to Treatment Period Month 2 | 92.73 (261.37) | -25.52 (49.62)
  Baseline to Treatment Period Month 3 | 114.10 (354.77) | 73.42 (224.71)

6. Secondary Outcome: Headache Days With Greater Than 50% Reduction
Description: Number of subjects with at least a 50% reduction in number of headache days reported in Baseline versus Treatment period Months 1, 2, and 3 in Sumatriptan/Naproxen Sodium arm vs. Naproxen Sodium arm.
Time Frame: Baseline Period collected at Day 31, Treatment Period Months 1, 2, and 3 collected at Days 61, 91, and 121.
Measure: Number; unit: participants
Arm/Group | Sumatriptan/Naproxen Sodium | Naproxen Sodium
Number analyzed (Participants) | 18 | 14
participants
  Baseline to Treatment Period Month 1 | 1 | 3
  Baseline to Treatment Period Month 2 | 2 | 3
  Baseline to Treatment Period Month 3 | 3 | 6

7. Secondary Outcome: Migraine Attacks With 50% Reduction
Description: Number of subjects with at least a 50% reduction in number of migraine attacks reported in Baseline versus Treatment period Months 1, 2, and 3 in Sumatriptan/Naproxen Sodium arm vs. Naproxen Sodium arm
Time Frame: Baseline Period collected at Day 31, Treatment Period Months 1, 2, and 3 collected at Days 61, 91, and 121.
Measure: Number; unit: participants
Arm/Group | Sumatriptan/Naproxen Sodium | Naproxen Sodium
Number analyzed (Participants) | 18 | 14
participants
  Baseline to Treatment Period Month 1 | 3 | 1
  Baseline to Treatment Period Month 2 | 2 | 0
  Baseline to Treatment Period Month 3 | 4 | 6

8. Secondary Outcome: Doses of Study Medication
Description: Total number of doses of study medication reported taken per participant in Treatment Period Months 1, 2, and 3 in Sumatriptan/Naproxen Sodium arm vs. Naproxen Sodium arm.
Time Frame: Treatment Period Months 1, 2, and 3 collected at Days 61, 91, and 121.
Measure: Mean (Standard Deviation); unit: doses of study medication
Arm/Group | Sumatriptan/Naproxen Sodium | Naproxen Sodium
Number analyzed (Participants) | 18 | 14
doses of study medication
  Treatment Period Month 1 | 11.00 (3.94) | 9.36 (5.53)
  Treatment Period Month 2 | 10.28 (6.39) | 8.86 (5.17)
  Treatment Period Month 3 | 10.28 (7.08) | 8.50 (6.04)

9. Secondary Outcome: Percent Change of Doses of Study Medication
Description: % change in number of doses during Baseline of triptans (Group A) and non-steroidal anti-inflammatory drugs(NSAIDs) (Group B) vs. doses during Treatment Period Months 1, 2, and 3 of study medication in the Sumatriptan/Naproxen Sodium arm vs. Naproxen Sodium arm. e.g.,Percent change=[(number of doses during Treatment Period Month 3 (Days 91-120)- number of doses during Baseline (Days 1-30)/number of doses during Baseline (Days 1-30)]*100%). The total number of subjects used in this analysis is different than the total number of subjects as the analysis is only looking at those subjects that were taking one of the study medications during Baseline.
Time Frame: Treatment Period Months 1, 2, and 3 collected at Days 61, 91, and 121.
Population: 12 Subjects did not take any triptans (Group A) or NSAIDs (Group B) during Baseline Period and were not included in Matched Pairs analysis of study medication taken.
Measure: Mean (Standard Deviation); unit: percent change of study medication
Arm/Group | Sumatriptan/Naproxen Sodium | Naproxen Sodium
Number analyzed (Participants) | 11 | 9
percent change of study medication
  Baseline to Treatment Period Month 1 | 130.8 (240.8) | 160.8 (399.2)
  Baseline to Treatment Period Month 2 | 114.9 (197.1) | 76.4 (152.5)
  Baseline to Treatment Period Month 3 | 96.1 (208.0) | 112.7 (228.0)

10. Secondary Outcome: Migraine Disability Assessment Test (MIDAS)
Description: Change in MIDAS total score from end of Baseline (Day 31) to end Treatment Period month 3 (Day 121) in the Sumatriptan/Naproxen Sodium arm vs. Naproxen Sodium arm.
  Total score of disability ranges:
  * 0 to 5, MIDAS Grade I, Little or no disability
  * 6 to 10, MIDAS Grade II, Mild disability
  * 11 to 20, MIDAS Grade III, Moderate disability
  * 21+, MIDAS Grade IV, Severe disability No subscales are present.
Time Frame: Baseline MIDAS collected at Day 31, Post final dose study medication MIDAS collected at Day 121.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Sumatriptan/Naproxen Sodium | Naproxen Sodium
Number analyzed (Participants) | 18 | 14
scores on a scale
  Baseline Day 31 | 28.7 (36.7) | 22.6 (21.6)
  Day 121 | 27.9 (20.3) | 24.1 (22.5)

11. Secondary Outcome: Compliance With Lifestyle Changes
Description: Self-assessed grade of compliance with lifestyle modification changes (where A=1, B=2, C=3, D=4, and F=5; lower scores represent better outcomes) in Sumatriptan/Naproxen Sodium arm vs. Naproxen Sodium arm.
Time Frame: Day 121
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Sumatriptan/Naproxen Sodium | Naproxen Sodium
Number analyzed (Participants) | 18 | 14
scores on a scale | 2.33 (0.69) | 2.43 (0.76)

12. Secondary Outcome: Percent Change in Headache Days All Treatment Periods Compared to Baseline
Description: Comparing the number of migraine headache days during Baseline Period Days 1-30 to number or migraine headache days reported in Treatment Period Month 1 (Days 31-60), Treatment Period Month 2 (Days 61-90), and Treatment Period Month 3 (Days 91-120) in Sumatriptan/Naproxen Sodium arm vs. Naproxen Sodium arm. e.g., Percent change=[ (total headache days during Treatment Period Month 3 (Days 91-120)-total headache days during Baseline (Days 1-30)/total headache days during Baseline (Days 1-30)]*100%).
Time Frame: Baseline Period collected at Day 31, Treatment Period Months 1, 2, and 3 collected at Days 61, 91, and 121.
Measure: Mean (Standard Deviation); unit: percent change of migraine headache days
Arm/Group | Sumatriptan/Naproxen Sodium | Naproxen Sodium
Number analyzed (Participants) | 18 | 14
percent change of migraine headache days
  Baseline to Treatment Period Month 1 | -1.70 (37.94) | -26.86 (31.74)
  Baseline to Treatment Period Month 2 | -4.39 (43.66) | -21.44 (28.79)
  Baseline to Treatment Period Month 3 | -13.50 (34.80) | -36.50 (36.48)

ADVERSE EVENTS:
Arm/Group | Sumatriptan/Naproxen Sodium | Naproxen Sodium
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/20
Other Adverse Events (participants affected / at risk) | 5/19 | 6/20
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sumatriptan/Naproxen Sodium (N=19) | Naproxen Sodium (N=20)
Allergic Rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Allodynia (Nervous system disorders) | 1 (82) | 0 (0) — Allodynia reported by one patient for 2 hours after every administration of study medication.
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Fever (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0)
Kidney Stone Pain Flare (Renal and urinary disorders) | 0 (0) | 1 (1)
Left Arm Numbness (Nervous system disorders) | 0 (0) | 1 (1)
Left Arm Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Left Hand Numbness (Nervous system disorders) | 0 (0) | 1 (1)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Right Chest Wall Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Root Canal Pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (2)
Stiffness in neck (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Weight Gain (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Wisdom Teeth Extraction Pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less